CLINICAL TRIAL: NCT04520568
Title: Preventing Deoxygenation With High Flow Nasal Cannula Oxygen During Sedation for Video-assisted Thoracoscopic Surgery: A Randomized Controlled Trial
Brief Title: High Flow Nasal Cannula Oxygen During Sedation for Video-assisted Thoracoscopic Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, rehab zayed, Assisstant Professor of Anesthesia, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 0304712
Record Dates: First submitted 2020-08-16; First posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Chronic Obstructive Pulmonary Disease; Respiratory Failure
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HFNC group (Active Comparator): For HFNC group, F&P AIRVOTM 2 will be adjusted to give the patients the oxygen flow at 50L/min and the FiO2 at 1.0.Then after three minutes of preoxygenation, sedation will be conducted by giving 25 µg fentanyl and a bolus of 1 mg/kg propofol followed by continuous infusion of propofol using a target-controlled infusion system (TCI pump TE371; Terumo Corporation, TokyoJapan).
  Interventions: Combination Product: High flow nasal cannula
- control group (Placebo Comparator): induction of general anaesthesia will be done using 2 mg/kg propofol and 1 µg/kg fentanyl. Double lumen tube will be facilitated by cisatracurium 0.2 mg/kg. Anaesthesia will be maintained with isoflurane 0.8 %-1% in 100% oxygen and maintenance dose of cisatracurium 0.02 mg/kg when needed. At the end of surgery, residual neuromuscular paralysis will be antagonized with neostigmine 0.05 mg/kg and atropine 0.01 mg/kg.
  Interventions: Combination Product: CONTROL

INTERVENTIONS:
Combination Product: High flow nasal cannula — using sedation with the HFNC F&P AIRVOTM 2 to maintain oxygenation
  Other Names: HFNC
  Arms: HFNC group
Combination Product: CONTROL — using general anaesthesia with one lung ventilation (OLV) technique
  Arms: control group

SUMMARY:
High-flow nasal cannula (HFNC) is a device that delivers10 to 70 L min-1 of heated, humidified 100% oxygen via nasal route. It provides positive airway pressure, decreases dyspnea, decreases the work of breathing, and improves comfort

DETAILED DESCRIPTION:
Beneficial effects of the HFNC system have been assessed based on 3 physiologic conditions: decreased dead space, a high concentration of inspiratory oxygen, and positive pressure in the oro-laryngeal cavity.Studies have shown that it improves oxygenation in various perioperative settings such as the apneic patients, patients with respiratory failure , and patients undergoing bronchoscopy

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status II and III,
* undergoing VATS

Exclusion Criteria:

* refusal of patients
* extrem of age

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-11-10 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
arterial partial pressures of oxygen | two hours
  an arterial blood sample will be taken after induction of anaesthesia then every 10 min till the end of the operation.
pH measurement | two hours
  an arterial blood sample will be taken after induction of anaesthesia then every 10 min till the end of the operation.

CONTACTS AND LOCATIONS:
Overall Officials: Rehab A. Abd Elaziz, Ass.Prof., Principal Investigator — Alexandria University
Locations (1):
- Rehab Abd Elraof Abd Elaziz, Alexandria, Egypt